CLINICAL TRIAL: NCT00473928
Title: Assessment of Safety of Intravitreal POT-4 Therapy for Patients With Neovascular Age-Related Macular Degeneration (AMD)
Brief Title: Safety of Intravitreal POT-4 Therapy for Patients With Neovascular Age-Related Macular Degeneration (AMD)
Acronym: ASaP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Potentia Pharmaceuticals, Inc. (Industry)
Responsible Party: Clinical Research Director, Potentia Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: POT-CP1006
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Age-Related Macular Degeneration
Keywords: Macular; degeration; Complement
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: POT-4 — Single intravitreal injection.

SUMMARY:
The objective of this study is to provide initial safety and tolerability information of intravitreal POT-4 for treatment of patients with AMD

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the leading cause of blindness for individuals over fifty-five years of age that live in the industrialized world. It affects 5-10 million people in the US and as many as 30 million worldwide. There are two forms of the disease, both of which cause a loss of central vision. Approximately eighty-five percent of patients have the less severe dry form that produces gradual but rarely complete vision loss. The remaining fifteen percent have the severe wet, or exudative, form that causes rapid, disabling blindness. Wet AMD is further characterized by choroidal neovascularization (CNV), a growth under the macula of abnormal blood vessels originating from the choroidal capillary bed. Research has linked chronic inflammation to both forms of AMD.

Only recently, unrestrained complement activation was identified in genetic studies to be one of the key mechanisms in the pathogenesis of AMD. It has also been demonstrated that complement activation plays a crucial role in the development of CNV. Therefore, the use of intravitreal complement inhibitors may be beneficial in participants subjects with neovascular AMD.

This prospective, uncontrolled, non-randomized, dose-escalating, pilot Phase I study will provide initial safety and tolerability information on intravitreal complement inhibitor (POT-4) therapy in AMD patients with subfoveal CNV.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the IRB-approved informed consent document for the study.
* Age ≥ 50 years.
* In the study eye, diagnosis of exudative AMD defined by the presence of drusen larger than 63 μm.
* In the study eye, the presence of a choroidal neovascular lesion, either predominantly or minimally classic or occult with no classic in nature, determined by the Digital Angiography Reading Center (DARC) with the CNV defined by its fluorescein angiographic (FA) features.
* The lesion must contain some visible active CNV, but the active CNV need not be under the fovea itself.
* Visual acuity of 20/60 or worse in the study eye as measured on an ETDRS chart.
* Retinal photographs and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice, can be obtained.
* Willingness to comply with the protocol.

Exclusion Criteria:

* Choroidal neovascularization in the study eye associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis or posterior uveitis, etc.
* Decreased vision, in the study eye, due to retinal disease not attributable to CNV, such as nonexudative forms of AMD, geographic atrophy, inherited retinal dystrophy, uveitis or epiretinal membrane, a vitelliform-like lesion of the outer retina (e.g., as in pattern dystrophies or basal laminar drusen), idiopathic parafoveal telangiectasis, or central serous retinopathy. Participants who have any additional ocular diseases that have irreversibly compromised or, during follow-up, could likely compromise the VA of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
* Decreased vision, in the study eye, due to significant media opacity such as corneal disease or cataract, or opacity precluding photography of the retina.
* Cataract surgery within three months of enrolment.
* Presence of hemorrhage greater than 50% of the CNV lesion.
* Previous PDT treatment in the study eye (eye to be treated) within 30 days prior to enrollment in the study.
* Previous extrafoveal or juxtafoveal thermal laser photocoagulation in the study eye (eye to be treated) is allowed, if performed at least 30 days prior to enrollment in the study.
* Previous Macugen (pegaptanib) injection in the study eye (eye to be treated) within 30 days prior to enrollment in the study.
* Previous Lucentis (ranibizumab) injection in the study eye (eye to be treated) within 30 days prior to enrollment in the study.
* Previous Avastin (bevacizumab) injection in the study eye (eye to be treated) within 30 days prior to enrollment in the study.
* Previous corticosteroid injection in the study eye (eye to be treated) within 180 days prior to enrollment in the study.
* History of peribulbar corticosteroid injection within 6 months prior to the start of the trial.
* History of oral steroid use at any time during the 30 days prior to randomization.
* Intraocular surgery (including lens replacement surgery) within 6 weeks prior to randomization.
* Participation in any other clinical study or are receiving, or have received any experimental systemic treatment for AMD (e.g.: retinoic acid, thalidomide) or any other investigational new drug within 12 weeks prior to the start of study treatment.
* Medical problems that make consistent follow-up over the treatment period unlikely (e.g. stroke, severe MI, end stage malignancy), or in general a poor medical risk because of other systemic diseases or active uncontrolled infections.
* Advance coronary artery disease or cerebral vascular disease.
* Premenopausal women not using adequate contraception
* Pregnancy or lactation
* Hypersensitivity to Fluorescein

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Local and systemic assessments of participant safety. - Incidence and severity of ocular adverse events - Incidence and severity of non-ocular adverse events | Within 30 days after POT-4 administration

SECONDARY OUTCOMES:
Secondary outcomes will investigate the safety and further define the efficacy profile including changes in visual acuity, retinal thickening, and CNV lesion (size and composition). | For up to a year after POT-4 administration

CONTACTS AND LOCATIONS:
Overall Officials: Jason Slakter, MD, Principal Investigator — Potentia Pharmaceuticals
Locations (6):
- United States (6):
  - United States, Arizona, Tucson, Arizona
  - United States, California, Beverly Hills, California
  - United States, Florida, Gainesville, Florida
  - United States, Florida, Miami, Florida
  - United States, Minnesota, Rochester, Minnesota
  - United States, New Hampshire, Portsmouth, New Hampshire